CLINICAL TRIAL: NCT00139438
Title: Improving Management of Patients at High Risk for Osteoporotic Fractures
Brief Title: Improving Management of Patients at High Risk for Osteoporotic Fractures (0000-038)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 0000-038; 038; 2005_049
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

INTERVENTIONS:
Behavioral: Disease Management Assessment

SUMMARY:
The purpose of this study is to assess the impact of disease management interventions on percent receiving a bone densitometry test and percent appropriately prescribed a medication for osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Members of the Horizon Blue Cross Blue Shield of New Jersey who are at risk for osteoporosis based on age (women age 65 or older, men and women age 45 or older who have a history of fragility fracture or have a history of taking oral glucocorticoids over 3 months).

Exclusion Criteria:

* Individuals who are not members of Horizon Blue Cross Blue Shield of New Jersey and who otherwise do not meet the inclusion criteria.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4266
Dates: Start 2004-09; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
A composite measure of bone mineral density (BMD) testing and/or osteoporosis medications prescriptions.

SECONDARY OUTCOMES:
BMD testing, osteoporosis medication prescriptions, fracture

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H. Solomon, M.D., M.P.H., Principal Investigator — Brigham and Woman's Hospital